CLINICAL TRIAL: NCT05437731
Title: Evaluation of Titanium Mesh Coated With Natural Hydroxyapatite Nanocrystals in Orbital Reconstruction (Randomized Controlled Clinical Trial)
Brief Title: Titanium Mesh Coated With Natural Hydroxyapatite Nanocrystals in Orbital Reconstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Orbital_Reconstruction_2022
Record Dates: First submitted 2022-06-27; First posted 2022-06-29 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Orbital Deformity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental)
  Interventions: Other: Coated titanium mesh
- Control group (Active Comparator)
  Interventions: Other: Uncoated titanium mesh

INTERVENTIONS:
Other: Coated titanium mesh — patients will undergo repairing of defects or reconstruction using the titanium mesh coated with hydroxyapatite nanocrystals.
  Arms: Study group
Other: Uncoated titanium mesh — patients will undergo reconstruction using the conventional uncoated titanium mesh.
  Arms: Control group

SUMMARY:
Reconstruction of maxillofacial continuity defects has always been a challenging task for scientists and surgeons over the years. The main goal of the reconstruction of the maxillofacial region is to restore facial form, function, and full rehabilitation of occlusion and articulation. A refinement in surgical technique and methods of reconstruction has improved patients' quality of life. Aim of this study: Evaluation of titanium mesh coated with natural hydroxyapatite in orbital reconstruction.

DETAILED DESCRIPTION:
Twelve patients having orbital defects will be selected. Six defects will be reconstructed using titanium mesh coated with natural hydroxyapatite nanocrystals (study group) and the other six will be treated with uncoated titanium mesh (control group). Patients will be evaluated clinically, then a radiographic follow-up will be performed immediately postoperatively and after three months to evaluate the bone density at the defect. Also, the coated and uncoated titanium mesh will be mechanically evaluated to compare the tensile strength of the two groups.

ELIGIBILITY:
Inclusion Criteria:

* All patients requiring reconstruction of acquired orbital defects using titanium mesh.
* Both genders with age group ranging from 18-60 years old.
* Limited size defects according to Cordeiro and Santamaria.
* Isolated unilateral or bilateral orbital fractures or combined with other facial fractures.
* Orbital reconstruction after removal of benign pathological lesions.

Exclusion Criteria:

* Infected fracture sites.
* Chronic systemic diseases such as uncontrolled diabetes, rheumatoid arthritis, metabolic bone disease, immunocompromised status etc.
* Defects requiring soft tissue reconstruction.
* Patients suffering from burns.
* Patients suffering from carcinomas and sarcomas in the oral cavity.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-10-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Change in wound healing criteria | after 24-hours, one week, four weeks, and six weeks
  The sutured wounds will be examined for signs and symptoms of infection. Yes: for presence of signs and sympotms No: for absence of signs and symptoms
Change in bone density | at baseline and 3 months
  All patients will be radiographically examined immediately and 3 months postoperatively using multi-slice computerized tomography (CT) using OnDemand3D software

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Clinic of Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Alexandria University, Alexandria, Egypt